CLINICAL TRIAL: NCT06007495
Title: Pilot Physiological Evaluation of an Investigational Mask with Expiratory Washout.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIP_336
Record Dates: First submitted 2023-08-14; First posted 2023-08-23 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-09

CONDITIONS: Acute Hypercapnic Respiratory Failure; Acute Hypoxemic Respiratory Failure
Keywords: Non-invasive Ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Randomized Cross-Over study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Single-limb non-invasive ventilation with expiratory washout (Experimental): In a random order, 30 minute period of non-invasive ventilation using the investigational mask, a vented full-face mask with expiratory washout
  Interventions: Device: Investigational full-face mask with expiratory washout
- Single-limb non-invasive ventilation (Active Comparator): In a random order, 30 minute period of non-invasive ventilation with a conventional vented full-face mask (RT077 or equivalent)
  Interventions: Device: Conventional full-face mask - single-limb
- Dual-limb non-invasive ventilation (Active Comparator): In a random order, 30 minute period of non-invasive ventilation with a conventional vented full-face mask (RT076 or equivalent)
  Interventions: Device: Conventional full-face mask - dual-limb

INTERVENTIONS:
Device: Investigational full-face mask with expiratory washout — With cross-over in randomized order, mask worn for 30 minutes with prescribed single-limb non-invasive ventilation
  Arms: Single-limb non-invasive ventilation with expiratory washout
Device: Conventional full-face mask - single-limb — With cross-over in randomized order, conventional mask such as RT077, worn for 30 minutes with prescribed single-limb non-invasive ventilation
  Other Names: RT077
  Arms: Single-limb non-invasive ventilation
Device: Conventional full-face mask - dual-limb — With cross-over in randomized order, conventional mask such as RT076, worn for 30 minutes with prescribed dual-limb non-invasive ventilation
  Other Names: RT076
  Arms: Dual-limb non-invasive ventilation

SUMMARY:
The goal of this pilot randomized cross-over study is to compare the effect of a full-face mask with expiratory washout to a conventional full face mask on non-invasive ventilation (NIV) in patients with acute hypercapnic, and acute hypoxemic, respiratory failure. The main questions it aims to answer are:

* Does a mask with expiratory washout improve minute ventilation in patients using non-invasive ventilation compared with a conventional single-limb NIV mask
* How does a mask with expiratory washout affect respiratory variables compared with a dual-limb NIV mask.

Participants already prescribed NIV will undergo 3 arms of the investigation in a randomized order:

* Single-limb NIV with investigation mask (with expiratory washout)
* Single-limb NIV with conventional mask
* Dual-limb NIV with conventional mask

DETAILED DESCRIPTION:
The investigational mask has been designed to deliver non-invasive ventilation (NIV) therapy with expiratory washout.

Expiratory washout is a technique designed to flush the upper airway of carbon dioxide at the end of expiration. During conventional NIV the gas at end of exhalation contributes to the functional dead space and "wasted" ventilation. The primary purpose of expiratory washout is to flush the upper airway with fresh gas during exhalation so the next supported breath which drives gas back into the alveolar regions has reduced carbon dioxide.

Patients that are admitted to hospital with acute (hypercapnic or hypoxemic) respiratory failure, as assessed by normal hospital protocols, and starting or prescribed to start NIV therapy will be considered for the investigation. Once stabilized on NIV by the physician in charge of their care, eligible patients will be assessed against the inclusion/exclusion criteria and enrolled into the study if applicable.

Participants that are enrolled into the study will be put onto oxygen therapy via nasal cannula for 15 minutes, during which time baseline measurements of physiological parameters (such as respiratory rate, tidal volume, minute ventilation and blood gases) and dyspnea scores will be recorded.

Following baseline measurements, 32 participants will be randomized into one of the 3 investigational arms and receive NIV with heated humidification according to the randomization protocol for 30 minutes each arm (90 minutes total). The same measurements will be recorded at the end of each 30-minute investigational arm. Participants will cross over to the other 2 conditions consecutively in a random order, each for 30 minutes.

The ventilator settings (press support ventilation (PSV), positive end expiratory pressure (PEEP)) will be the following: PSV for tidal volume comprised between 6 and 8 millilitres per kilogram (ml/kg) predicted body weight (PBW), a titration period will be planned at the beginning of the first study period to target a tidal volume of 7 +/-1 ml/kg PBW and the PSV level will be kept constant thereafter. PEEP will be set according to the physician in charge (between 5 and 10 centimetres of water (cmH2O)) if NIV was used before inclusion or will be set by the investigators between 5 and 10 cmH2O. The fraction of inspired oxygen will be titrated manually to target peripheral saturation of oxygen of 88-92% in patients with hypercapnia and 90-94% in patients without hypercapnia.

Once the investigation is complete, and participants have successfully finished all 3 arms of NIV therapy, the standard NIV protocols as per local hospital will resume, and participants will return to the care of their usual physician.

ELIGIBILITY:
Inclusion Criteria:

* No indication of intubation upon evaluation by physician in the next 2 hours
* Fits the investigational mask

Specific for hypercapnic patients 1 of the following criteria

* Patients hospitalized with acute respiratory failure (ARF) stabilized and tolerating NIV or;
* Patient admitted to hospital with ARF with one criteria for NIV among the following:

  * Acute hypercapnic respiratory failure with hypercapnia and acidosis (Partial pressure of arterial carbon dioxide (PaCO2) > 45 millimeters of mercury (mmHg) and pH < 7.38) or
  * Post-extubation period within 48 hours, in patients with high risk of re-intubation

Specific for hypoxemic patients

1 of the following criteria

* Hypoxemic respiratory failure without hypercapnia requiring nasal high flow or;
* Hypoxemic respiratory failure without hypercapnia requiring NIV or;
* Conventional oxygen therapy (COT) > 6 liters per minute (L/min) with peripheral oxygen saturation (SpO2) < 92%

Exclusion Criteria:

* Refusal to participate in the study
* Inability to provide informed consent
* Infectious isolation
* Facial deformity, burns or morphology that prevents adequate mask placement
* Claustrophobia
* Nausea
* Presence of nasogastric tube
* Pneumothorax
* Confusion or loss of consciousness
* Severe upper gastro-intestinal bleeding
* Any other condition, which at the investigators discretion, is believed may present a safety risk or impact the feasibility of the study or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Minute Ventilation | Recorded at baseline and the end of each 30-minute period of non-invasive ventilation over 1 hour and 30 minutes of data measurement
  Variations of the minute ventilation in the three different arms (Investigational mask, single-limb conventional, dual-limb conventional)

SECONDARY OUTCOMES:
Tidal Volume | Recorded at baseline and the end of each 30-minute period of non-invasive ventilation over 1 hour and 30 minutes of data measurement
  Changes in tidal volume over the three different arms
Respiratory Rate | Recorded at baseline and the end of each 30-minute period of non-invasive ventilation over 1 hour and 30 minutes of data measurement
  Changes in respiratory rate over the three different arms
Blood gases | Recorded at baseline and the end of each 30-minute period of non-invasive ventilation over 1 hour and 30 minutes of data measurement
  Changes in blood gas values over the three different arms
Dyspnoea Score | Recorded at baseline and the end of each 30-minute period of non-invasive ventilation over 1 hour and 30 minutes of data measurement
  Changes in dyspnea score over the three different arms. Dyspnea measured with the modified Borg dyspnea score, which utilizes a scale of 0 to 10 where 0 represents no dyspnea and 10 represents maximal dyspnea.
Mask Comfort Score | Recorded at baseline and the end of each 30-minute period of non-invasive ventilation over 1 hour and 30 minutes of data measurement
  Changes in mask comfort score over the three different arms. Mask comfort will be measured with a subjective likert scale of comfort where 1 represents maximal comfort, and 5 represents least comfort.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Quebec